CLINICAL TRIAL: NCT07381699
Title: MRG003 Combined With Pucotenlimab as First-Line Therapy for Recurrent/Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial
Brief Title: MRG003 Combined With Immunotherapy in Recurrent/Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, Director of head and neck oncology Department, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH-2026-NPC-PII-001-MRG003
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Recurrent/Metastatic Nasopharyngeal Carcinoma
Keywords: Recurrent/Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRG003 + PD-1 inhibitor (Experimental)
  Interventions: Drug: MRG003 and Pucotenlimab

INTERVENTIONS:
Drug: MRG003 and Pucotenlimab — MRG003 combined with Pucotenlimab, administered on Day 1 every 3 weeks (D1 Q3W), until disease progression (PD), unacceptable toxicity, or death.

SUMMARY:
This study was designed to compare the efficacy and safety of MRG003 combined with Pucotenlimab as first-line treatment for recurrent or metastatic nasopharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Life expectancy ≥ 3 months.
4. Histologically or cytologically confirmed nasopharyngeal carcinoma (NPC).
5. Metastatic NPC (Stage IVB, AJCC 8th) or locally recurrent NPC unfit for curative local therapy (e.g., surgery, TACE, radiotherapy).
6. Must be treatment-naive for recurrent or metastatic NPC.
7. Must have ≥ 1 measurable lesions as defined per RECIST v1.1.
8. Adequate organ function.
9. For women of childbearing potential: negative pregnancy test within 7 days prior to treatment initiation. All participants of childbearing potential must agree to use effective contraception during the study and for 1 year after treatment discontinuation.
10. Willing and able to provide written informed consent and comply with study procedures and follow-up visits.

Exclusion Criteria:

1. Peripheral neuropathy of Grade 2 or higher.
2. Anticipated need for any other local or systemic anti-tumor therapy during the study period.
3. Diagnosed and/or treated additional malignancy within 5 years of enrollment, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, and/or curatively-resected in situ cervical and/or breast carcinoma.
4. Active central nervous system (CNS) metastases or carcinomatous meningitis.
5. Laboratory values within 7 days prior to enrollment falling outside specified eligibility ranges (e.g., Child-Pugh C; creatinine clearance <30 mL/min; serum sodium <135 mmol/L; serum potassium <3.5 mmol/L).
6. Severe or uncontrolled cardiovascular disease.
7. History of or current interstitial lung disease, severe chronic obstructive pulmonary disease with respiratory failure, severe pulmonary insufficiency, or symptomatic bronchospasm.
8. Active infection requiring systemic therapy.
9. Severe, or uncontrolled systematic diseases (e.g., uncontrolled hypertension, or uncontrolled diabetes).
10. Known history of testing positive for human immunodeficiency virus (HIV).
11. Known history of allogeneic hematopoietic stem cell, bone marrow, or solid organ transplantation.
12. Known active hepatitis B or C infection, or other severe liver disease.
13. Live vaccine within 30 days prior to the first dose.
14. Residual toxicity from prior anti-tumor therapy higher than grade 1 (except alopecia, fatigue, and grade 2 hypothyroidism).
15. Active autoimmune disease or a history of autoimmune disease requiring systemic steroid or immunosuppressive therapy. The following conditions are not exclusionary: mild asthma controlled with intermittent bronchodilators; stable hypothyroidism on hormone replacement; vitiligo; Graves' disease; or Hashimoto's disease.
16. Known history of Grade 3 or higher hypersensitivity to any component of MRG003 or to other monoclonal antibodies.
17. Uncontrolled pleural effusion, ascites, or pericardial effusion.
18. Pregnancy, breastfeeding, or unwillingness to use a highly effective method of contraception during the treatment period and for at least 180 days after the last dose.
19. Any other condition that, in the opinion of the investigator, may compromise the safety and integrity of the study participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 2 years.
  Defined as the period from treatment initiation until disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years.
  Defined as the proportion of patients whose tumors shrink to complete response (CR) or partial response (PR) and remain for a certain period of time according to RECIST 1.1.
Disease Control Rates (DCR) | Up to approximately 2 years.
  Defined as the proportion of subjects who achieve CR+PR+stable disease (SD) for a certain period of time according to RECIST 1.1.
Duration of Response (DoR) | Up to approximately 2 years.
  Defined as the time from the first assessment of CR and PR to the first assessment of PD or death caused by any cause according to RECIST 1.1.
Overall Survival (OS) | Up to approximately 2 years.
  Defined as the period from treatment initiation until death from any cause.
Adverse events | Up to approximately 2 years.
  NCI-CTCAE 5.0 standard was adopted, and the safety was assessed mainly by ECOG-PS score, physical examination, clinical laboratory tests, electrocardiogram, and adverse event results.

IPD SHARING:
Plan to Share IPD: Undecided